CLINICAL TRIAL: NCT05046223
Title: Analysis of Intraoperative Homeostasis and Postoperative Recovery After Interventional Bronchoscopy With Different Anesthetic Management
Brief Title: Comparison of iGel and THRIVE on Bronchoscopic Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 202011092RINA
Record Dates: First submitted 2021-08-13; First posted 2021-09-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Lung Diseases; Total Intravenous Anesthesia; Tracheal Diseases
MeSH Terms: conditions — Lung Diseases; Tracheal Diseases | interventions — Cryotherapy; Hemodynamics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high-flow nasal oxygen (Experimental): THRIVE( Transnasal humidified rapid-insufflation ventilatory exchange), a method of high-flow nasal oxygen (HFNO), is planned to applied for bronchoscopic interventions
  Interventions: Procedure: The responses to bronchoscopic insertion for bronchoscopic interventions such asTBNA, Cryotherapy, etc.; Procedure: postoperative recovery
- supraglottic devise (Active Comparator): iGel, a supraglottic devise with tip in upper esophagus, is planned to applied for bronchoscopic interventions
  Interventions: Procedure: The responses to bronchoscopic insertion for bronchoscopic interventions such asTBNA, Cryotherapy, etc.; Procedure: postoperative recovery

INTERVENTIONS:
Procedure: The responses to bronchoscopic insertion for bronchoscopic interventions such asTBNA, Cryotherapy, etc. — cough response, the changes of BP, HR, SpO2, Trans dermal CO2 during bronchoscopic interventions
  Other Names: hemodynamic and ventilatory responses from insertion of broncoscopy to the end of bronchoscopic interventions
Procedure: postoperative recovery — anesthetic recovery in postoperative care unit recovery of swallowing by questionnaire in POD1

SUMMARY:
THRIVE and iGEL were applied for maintain oxygenation in bronchoscopic interventions which could not performed with an endotracheal tube. However, besides the risk of desaturation, the differences on difficulties to approach vocal cords, the responses to spay of local anesthetics including cough or spasm, the CO2 elimination, the hemodynamic changes, and the effects on postoperative recovery are rarely investigated.

DETAILED DESCRIPTION:
THRIVE and iGEL were applied for maintain oxygenation in bronchoscopic interventions which could not performed with an endotracheal tube. Unlike the nasal cannula with THRIVE, the tips of iGel are located in upper esophagi, it may affect the postoperative swallowing, especially for the aged group. However, the bronchoscopic approach may be easier for an established route to vocal cords. With shared airway for ventilation and interventions, CO2 elimination is hardly monitored besides the risk of desaturation.

In this study, THRIVE or iGel was planned to be randomized used for bronchoscopic interventions in an adult group (age 20-65) and an aged group (age over 65). The difficulties to approach vocal cords, the responses to spay of local anesthetics including cough or spasm, the CO2 elimination, the hemodynamic changes, and the effects on postoperative recovery are compared between THRIVE and iGel groups.

ELIGIBILITY:
Inclusion Criteria:

* plan to receive bronchoscopic interventions with total intravenous anesthesia

Exclusion Criteria:

* awake bronchoscopy pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
difficulty of bronchoscopic approach | from bronchoscopic insertion to visualize vocal cords
  time from insertion to visualize vocal cord, records of manipulations if applied
response to spraying local anesthetics by bronchoscopy | from visualizng vocal cords to complete local anesthetic spray in trachea and main bronchi
  the status of vocal cords visualized (relaxed, closed, relaxed but close with spray of local anesthetics); cough scale during bronchoscopic insertion and spray of local anesthetics

SECONDARY OUTCOMES:
hemodynamic changes | from bronchoscopic insertion to 20 minutes after completion of local anesthetic spraying
  changes on MAP (mmHg)
cough scale | from bronchoscopic insertion to the end of procedure
  cough intensity X times
SPO2 | every 5 minutes from bronchoscopic insertion to the end of procedure
  pulse oximeter, hemoglobin saturation (%)
Transdermal CO2 | every 5 minutes from bronchoscopic insertion to the end of procedure
  data obyenied from transdermal CO2 (mmHg)
postanesthetic recovery | from admission to PACU to discharge from PACU
  time stay in postoperative care unit (minutes)

OTHER OUTCOMES:
EAT-10 questionnaire (score):0-40 | preoperative and postoperative day 1
  EAT-10 for postbronchoscopic swallowing dysfunction, from 0 (normal swallowing) to 40 (extreme difficulty on swallowing)

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Chang Tsai, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Cancer Center, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
if there is similar investigation
Supporting Information: CSR
Time Frame: 1 year after completion of investigation